CLINICAL TRIAL: NCT04680403
Title: Video Telehealth Exercise Training in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Stefanie Krick MD, MD, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-300006495; Vertex Innovation Award (Other: Vertex Pharmaceuticals)
Record Dates: First submitted 2020-12-17; First posted 2020-12-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- supervised exercise plan (Experimental): patients will receive a tailored exercise regimen and behavior change techniques focused on adherence to the exercise program. These will be delivered by using a video platform, much liker telehealth clinic appointments. These telehealth visits will be over a 12-week period, occur 3 times a week, and last for 1 hour each.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — supervised exercise paired with coaching on behavior change techniques over 12 weeks (3 weekly sessions) and will have monthly phone follow-ups and clinic follow-ups after 3 and 6 months.
  Other Names: Behavior Change Coaching

SUMMARY:
The purpose of this research study is to begin an exercise program for patients with a cystic fibrosis (CF) exacerbation.

DETAILED DESCRIPTION:
The study will enroll 25 patients with CF during an introduction visit and initiate an ambulatory 1) tailored exercise regimen and 2) behavior change techniques focused on adherence and sustainability of exercise. The intervention will be delivered via a data-enabled smartphone with video capabilities facilitating live and interactive two-way video-conferencing using a HIPAA compliant app. Participants will receive supervised exercise paired with coaching on behavior change techniques over 12 weeks in 3 weekly 1-hour sessions, and will have monthly phone follow-ups and clinic follow-ups at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

Diagnosed with Cystic Fibrosis 18 years old and older clinically stable with no exacerbation within 6 weeks

Exclusion Criteria:

any comorbidity that precludes exercise

-

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and acceptability | 6 months
  Feasibility and acceptability will include patients willingness to participate

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Krick, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No